CLINICAL TRIAL: NCT07109141
Title: Registry of Atrial Arrhythmia Ablation Procedures Using Pulsed Field Ablation in Poland
Acronym: PFA Registry
Status: Recruiting | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Stanisław Tubek, MD, PhD, Wroclaw Medical University
Other Study IDs: 435/2024
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation (AF); Atrial Flutter; Atrial Tachycardia; Ablation Techniques; Pulsed Field Ablation
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing PFA ablation of atrial arrythmia: All patients undergoing PFA ablation procedure of atrial arrythmia will be invited to enter the study.
  Interventions: Procedure: PFA ablation procedure of atrial arrythmia

INTERVENTIONS:
Procedure: PFA ablation procedure of atrial arrythmia — PFA ablation procedure of atrial arrythmia accroding to the particular patients needs

SUMMARY:
The aim of the described project is to establish a multicenter, nationwide registry of atrial arrhythmia ablation procedures using the Pulsed Field Ablation (PFA) method. These procedures have only recently begun to be performed in several centers across Poland. With proper coordination of the registry, this will enable the consolidation of clinical data and the expansion of knowledge regarding the efficacy and safety of these procedures.

DETAILED DESCRIPTION:
Background A relatively recent innovation in cardiac ablation is Pulsed Field Ablation (PFA), a technique based on the phenomenon of irreversible electroporation. This method is tissue-selective, affecting only myocardial cells. Clinical studies have confirmed the efficacy and safety of PFA in the treatment of paroxysmal atrial fibrillation (AF).

Although the catheters currently used for PFA are designed primarily for pulmonary vein isolation (PVI) in AF ablation, there are growing numbers of reports describing their successful application in the ablation of other arrhythmias-such as atrial flutter, atrial tachycardia, and even ventricular tachycardia. However, the efficacy of such procedures has not yet been systematically evaluated in experimental or clinical settings.

We believe that establishing a national registry documenting PFA procedures for atrial arrhythmias will provide valuable insights into the clinical efficacy, safety, and procedural techniques of this emerging treatment strategy. Furthermore, it will support the planning and design of future randomized clinical trials in this area.

Objectives The aim of the project is to establish a multicenter, nationwide registry of PFA-based ablation procedures for arrhythmias other than atrial fibrillation.

Study Design and Planned Procedures The project involves the collection of clinically relevant data from patients undergoing PFA procedures targeting arrhythmias outside the pulmonary veins.

Participation in the registry will not require any additional procedures during hospitalization beyond standard clinical care.

Patients will be followed for 12 months post-ablation. Follow-up will include telephone interviews conducted at 3, 6, and 12 months after the procedure. If necessary, based on the telephone assessment, patients may be invited for an in-person clinical evaluation at the center where the procedure was performed.

The registry will be coordinated by the Institute for Heart Diseases at the Jan Mikulicz-Radecki University Hospital in Wroclaw, Poland. Other hospitals in Poland performing PFA procedures will be invited to participate in the registry.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from the participant
* Subject is undergoing ablation of an atrial arrhythmia using the PFA

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lack of informed consent from the participant
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of supraventricular arrhythmia | 12 months
  Recurrence of any supraventricular arrhythmia recorded in the ECG and provided by the participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Department of Cardio, Jan Mikulicz Radecki University Hospital in Wroclaw, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided